CLINICAL TRIAL: NCT02454777
Title: High-Intensity Interval Training (HIT) for Breast Cancer Patients During Trastuzumab Use
Brief Title: High-Intensity Interval Training for Stage I-III Breast Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1B-14-5; NCI-2015-00579 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1B-14-5 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-05-21; First posted 2015-05-27 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM I (HIT group) (Experimental): Participants undergo HIT exercises over 30 minutes, thrice weekly for 8 weeks.
  Interventions: Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (Delayed group) (Active Comparator): Participants maintain their current sedentary activity level (< 60 minutes of total exercise per week) for 8 weeks. Participants document their weekly activity in an exercise log. Following completion of all study visits, participants are given the option to complete the HIT program as in Arm I.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Exercise Intervention — Undergo HIT
  Arms: ARM I (HIT group)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies the feasibility of high-intensity interval training in improving cardiovascular fitness in patients with stage I-III breast cancer undergoing chemotherapy with trastuzumab. Trastuzumab helps patients live longer, but may cause side effects to the heart. Aerobic exercise may help the heart function better, which may help protect it against side effects from trastuzumab. Exercise may also help reduce fatigue and prevent cancer from coming back. High-intensity interval training involves short bursts of higher intensity efforts with longer periods of recovery. This may also allow patients who cannot exercise for a long period of time to still be physically active. This trial studies whether patients can tolerate high-intensity interval training, and how well it works in improving fitness in patients with breast cancer receiving trastuzumab.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility (completion of > 80% exercise sessions) of utilizing high-intensity interval training (HIT).

II. To determine the effects of HIT on aerobic exercise adaptation when compared to delayed group.

III. To examine the effects of HIT on left ventricular function when compared to delayed group.

IV. To determine the effects of HIT on endothelial function, arterial stiffness, and vascular atherosclerosis when compared to delayed group.

OUTLINE: Participants are randomized to 1 of 2 groups.

ARM I: HIT (High-intensity Interval Training) group - Participants undergo HIT over 30 minutes, thrice weekly for 8 weeks.

ARM II: DEL (Delayed/usual care) group - Participants maintain their current sedentary activity level (< 60 minutes of total exercise per week) for 8 weeks. Participants document their weekly activity in an exercise log. Following completion of all study visits, participants are given the option to complete the HIT exercise program as in Arm I.

After completion of study, patients are followed up at weeks 9 and 17.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Diagnosed with early stage (I-III) breast cancer, without evidence of metastatic disease
* Planned (neo)adjuvant therapy with trastuzumab (Herceptin) and/or anthracycline-based chemotherapy
* Not currently pregnant or planning to become pregnant throughout the duration of cancer treatment
* Physician (oncologist) clearance to participate in exercise at moderate to high intensity
* Have read and signed study informed consent document (ICF)
* EXERCISE INCLUSION CRITERIA:
* Normal body temperature (=< 100 degrees F)
* Resting blood pressure and/or heart rate within normal limits
* Participants have not received intravenous or oral chemotherapy on the same day and prior to scheduled exercise session

Exclusion Criteria:

* Advanced stage (stage IV) or metastatic breast cancer diagnosis (screening for metastases with scans only needed if there is clinical suspicion for metastases)
* Medical history of coronary heart or artery disease, chronic or acute congestive heart failure or history of systolic or diastolic insufficiencies
* Uncontrolled hypertension or other uncontrolled chronic disease (e.g. diabetes mellitus, thyroid disease, pulmonary disease, etc.)
* Moderate to highly active level of physical activity (e.g. currently participating in >= 60 minutes of moderate aerobic activity weekly)
* Orthopedic or other restrictions or contraindications to high-intensity (cycling) exercise
* EXERCISE EXCLUSION CRITERIA:
* Presence of fever (>= 100 degrees F)
* Resting blood pressure and/or heart rate outside normal limits
* Participants have received intravenous or oral chemotherapy on the same day and prior to scheduled exercise session

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of utilizing HIT under clinical trial conditions, assessed using participant attendance rate | Up to 17 weeks
  The exercise program will be considered feasible if participants complete greater than 80% of exercise sessions. Participant attendance rates will be used to establish compliance and will be used to provide a perspective on how and to what extent cancer patients will participate in an experimental exercise intervention and what variations in exercise intensities may be tolerated. Feasibility will be assessed based on both program attendance as well as exercise time completed.

SECONDARY OUTCOMES:
Change in aerobic exercise adaptation measured by the maximum volume of oxygen uptake (VO2peak) (ml/kg/min) | Baseline to up to week 17
  A mixed-effect regression model will be fit to compare the mean changes in VO2peak (ml/kg/min) between groups. The effect of other covariates such as the menopausal age, severity of disease and the class of chemotherapy treatment and compliance rate on VO2peak (ml/kg/min) over time will also be examined.
Change in left ventricular function | Baseline to up to week 17
  A mixed-effect model will be fit to compare the mean changes in left ventricular ejection fraction, left ventricular end-diastolic volume, left ventricular end-systolic volume, and peak filling time. The effect of other covariates such as the menopausal age, severity of disease and the class of chemotherapy treatment and compliance rate on left ventricular function over time will also be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee K, Norris MK, Wang E, Dieli-Conwright CM. Effect of high-intensity interval training on patient-reported outcomes and physical function in women with breast cancer receiving anthracycline-based chemotherapy. Support Care Cancer. 2021 Nov;29(11):6863-6870. doi: 10.1007/s00520-021-06294-7. Epub 2021 May 20. PMID 34018031
- [Derived] Lee K, Kang I, Mack WJ, Mortimer J, Sattler F, Salem G, Dieli-Conwright CM. Feasibility of high intensity interval training in patients with breast Cancer undergoing anthracycline chemotherapy: a randomized pilot trial. BMC Cancer. 2019 Jul 3;19(1):653. doi: 10.1186/s12885-019-5887-7. PMID 31269914
- [Derived] Lee K, Kang I, Mack WJ, Mortimer J, Sattler F, Salem G, Lu J, Dieli-Conwright CM. Effects of high-intensity interval training on vascular endothelial function and vascular wall thickness in breast cancer patients receiving anthracycline-based chemotherapy: a randomized pilot study. Breast Cancer Res Treat. 2019 Sep;177(2):477-485. doi: 10.1007/s10549-019-05332-7. Epub 2019 Jun 24. PMID 31236810
- [Derived] Lee K, Kang I, Mortimer JE, Sattler F, Mack WJ, Fitzsimons LA, Salem G, Dieli-Conwright CM. Effects of high-intensity interval training on vascular function in breast cancer survivors undergoing anthracycline chemotherapy: design of a pilot study. BMJ Open. 2018 Jun 30;8(6):e022622. doi: 10.1136/bmjopen-2018-022622. PMID 29961039